CLINICAL TRIAL: NCT01004094
Title: Squire's Quest! II: Implementation Intentions and Children's FJV Consumption
Brief Title: Squire's Quest! II: Implementation Intentions and Children's Fruit, Juice, and Vegetable (FJV) Consumption
Acronym: SQ!II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Deborah Thompson, Associate Professor of Pediatrics, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Thompson_Squires_Quest_II; 5R01HD050595 (NIH)
Record Dates: First submitted 2009-10-28; First posted 2009-10-29 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Obesity; Cancer
Keywords: children; video games; internet; parents; fruit; vegetable; implementation intention; goal setting; fruit and vegetable consumption; obesity prevention; cancer prevention
MeSH Terms: conditions — Obesity; Neoplasms | interventions — Organizational Objectives

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- simple goal setting (Experimental): This group will only set a goal.
  Interventions: Behavioral: simple goal setting
- goal setting plus action intentions (Experimental): This group will set goals and form action intentions (plans) to facilitate goal attainment.
  Interventions: Behavioral: goal setting plus action intentions
- goal setting plus coping intentions (Experimental): This group will set goals and form coping intentions (plans) to facilitate goal attainment.
  Interventions: Behavioral: goal setting plus coping intentions
- goal setting plus action intentions plus coping intentions (Experimental): This group will set goals, form action intentions (plans), and form coping intentions (plans) to facilitate goal attainment.
  Interventions: Behavioral: goal setting plus action intentions plus coping intentions

INTERVENTIONS:
Behavioral: simple goal setting — This group will set goals only
  Other Names: goal setting
  Arms: simple goal setting
Behavioral: goal setting plus action intentions — This group will set goals and form action intentions (plans)
  Other Names: implementation intentions; action plans
  Arms: goal setting plus action intentions
Behavioral: goal setting plus coping intentions — This group will set goals and form coping intentions (plans)
  Other Names: implementation intentions; problem solving
  Arms: goal setting plus coping intentions
Behavioral: goal setting plus action intentions plus coping intentions — This group will set goals and form action intentions and coping intentions
  Other Names: implementation intentions; action plans; problem solving
  Arms: goal setting plus action intentions plus coping intentions

SUMMARY:
The primary purpose of this research is to test the effects of goal setting on fruit and vegetable goal attainment and consumption in a 10 episode video game. Factors associated with maintenance of behavior change will also be examined. Secondary purposes are to explore the impact of the intervention on psychosocial factors and the home environment. 400 parent-child pairs will be recruited for this research (800 participants total). Children will play the video game and participate in data collection activities. Parents will receive newsletters, have access to a healthy foods web site, and participate in data collection activities. A small subset will be randomly selected to participate in interviews about the intervention and its effect on the home food environment.

DETAILED DESCRIPTION:
Obesity is increasing among youth and is associated with increased risk of certain cancers and other chronic diseases. Fruit, juice, and vegetable (FJV) intake is associated with decreased risk of many types of cancer and obesity, but is well below the recommended minimum of five servings a day. Innovative methods are needed to promote increased consumption among youth.

Goal setting enhances goal attainment and, therefore, facilitates behavior change. Little research has been conducted, however, on the most effective goal setting methods to use with youth. Among adults, the formation of implementation intentions (a detailed plan of when, where, and how goals will be achieved) has been shown to enhance goal attainment and/or behavior change, including dietary change. Research is needed to determine if extending the goal setting process to include implementation intentions is an effective method for enhancing goal attainment, and therefore, increasing FJV intake among youth.

Squire's Quest! is a proven-effective 10-session, 5 week interactive multi media program that enabled children to increase FJV consumption by 1.0 servings a day. Total consumption was still well below five servings a day, however. Additionally, goal attainment was related to FJV consumption among certain sub-groups of youth. Therefore, additional work in this area is warranted. The research outlined in this proposal will expand the goal setting component of this successful intervention to include the formation of implementation intentions. Hypotheses related to the impact of implementation intentions on goal attainment and FJV consumption will then be tested. Issues related to maintenance of youth dietary behavior change will also be explored.

This project is relevant to public health because enhancing our understanding of how to more effectively help young children set and achieve FJV goals should result in increased FJV consumption, which should decrease risk of both obesity and certain cancers in a vulnerable segment of the population.

ELIGIBILITY:
Inclusion Criteria:

* child: 4th or 5th grade children who speak, write, and understand English; have access to a computer with high speed internet; provide written parental consent and child assent; and have a parent who speaks and understands English or Spanish who is willing to participate in the study
* Parents: parent or legal guardian of a child participating in the study

Exclusion Criteria:

* child: not meeting inclusion criteria; having physical, mental, or medical limitations that inhibit ability to fully participate in the study (answer questions online and over the phone, play the video game, eat fruit and vegetables); and/or not having a parent/legal guardian willing to participate in data collection activities.
* Parents. Exclusion criteria are limited to not meeting the inclusion criteria.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 800 (Actual)
Dates: Start 2009-10; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Fruit and vegetable consumption | baseline, immediate post, 3 months later

SECONDARY OUTCOMES:
Goal attainment | during intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- [Derived] DeSmet A, Liu Y, De Bourdeaudhuij I, Baranowski T, Thompson D. The effectiveness of asking behaviors among 9-11 year-old children in increasing home availability and children's intake of fruit and vegetables: results from the Squire's Quest II self-regulation game intervention. Int J Behav Nutr Phys Act. 2017 Apr 21;14(1):51. doi: 10.1186/s12966-017-0506-y. PMID 28431547
- [Derived] Thompson D, Ferry RJ Jr, Cullen KW, Liu Y. Improvement in Fruit and Vegetable Consumption Associated with More Favorable Energy Density and Nutrient and Food Group Intake, but not Kilocalories. J Acad Nutr Diet. 2016 Sep;116(9):1443-1449. doi: 10.1016/j.jand.2016.05.002. Epub 2016 Jun 15. PMID 27316780
- [Derived] Thompson D, Bhatt R, Vazquez I, Cullen KW, Baranowski J, Baranowski T, Liu Y. Creating action plans in a serious video game increases and maintains child fruit-vegetable intake: a randomized controlled trial. Int J Behav Nutr Phys Act. 2015 Mar 18;12:39. doi: 10.1186/s12966-015-0199-z. PMID 25890060
- [Derived] Thompson D, Bhatt R, Lazarus M, Cullen K, Baranowski J, Baranowski T. A Serious Video Game to Increase Fruit and Vegetable Consumption Among Elementary Aged Youth (Squire's Quest! II): Rationale, Design, and Methods. JMIR Res Protoc. 2012 Nov 21;1(2):e19. doi: 10.2196/resprot.2348. PMID 23612366